CLINICAL TRIAL: NCT03176082
Title: Mailed Reminders Plus Fecal Immunochemical Testing (FIT) to Increase Colorectal Cancer Screening Among Medicaid Beneficiaries in Mecklenburg County
Brief Title: Mailed Reminders Plus Fecal Immunochemical Testing
Acronym: MFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 16-0875
Record Dates: First submitted 2017-05-05; First posted 2017-06-05 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Cancer Screening; Colorectal Cancer
Keywords: colorectal cancer screening; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group will receive:
  1. A reminder letter indicating need for screening
  2. A FIT kit with completion instructions
  3. A health information card including the ability to update records for current screening and opt out from colon cancer screening communication from the Mecklenburg County Public Health Department (MCPHD)
  4. A pre-paid return mailer for FIT Kit
  Interventions: Other: Mailed Reminders with Fecal Immunochemical Testing kits
- Comparison Group (Active Comparator): Comparison group will receive:
  1. A reminder letter indicating need for screening
  2. Instructions for obtaining a FIT kit
  3. A health information card including the ability to update records for current screening and opt out from colon cancer screening communication from the MCPHD
  Interventions: Other: Reminder letter only

INTERVENTIONS:
Other: Mailed Reminders with Fecal Immunochemical Testing kits
  Arms: Intervention Group
Other: Reminder letter only
  Arms: Comparison Group

SUMMARY:
Purpose: The investigators propose to test the effectiveness, feasibility, and cost-effectiveness of a mailed reminder with and without FIT kits in a population of Medicaid enrollees in Mecklenburg County.

DETAILED DESCRIPTION:
Purpose: The investigators propose to test the effectiveness, feasibility, and cost-effectiveness of a mailed reminder with and without FIT kits in a population of Medicaid enrollees in Mecklenburg County.

Participants: Medicaid beneficiaries who are enrolled in Community Care of North Carolina, ages 52-64, currently living in Mecklenburg County, at average risk for colorectal cancer (CRC), with no record of recent CRC screening (FOBT within 12 months, colonoscopy within 10 years).

Procedures (methods): Participants will be identified through the state Medicaid database and randomized to receive either: 1) a mailed reminder to complete CRC screening including a FIT kit, instructions for completion, and a return mailer, OR 2) a mailed reminder to complete CRC screening only.

Any recipients testing positive will be guided by care managers from Community Care of North Carolina to ensure a follow-up colonoscopy is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Current Medicaid beneficiary,
2. Enrolled in Community Care Partners of Greater Mecklenburg (CCPGM),
3. 52-64 years old,
4. English or Spanish speaking,
5. No record of FOBT/FIT within 12 months or colonoscopy with 10 years, sigmoidoscopy within 5 years; barium enema within 5 years, CT colonography within 10 years,
6. No record of any CRC diagnosis or total colectomy

Exclusion Criteria:

1. < 52 or >64 years of age;
2. History of colorectal cancer or total colectomy (see attached table for codes),
3. Persons dually enrolled in Medicare,
4. Not enrolled in CCPGM, 5. Received FOBT or FIT within 12 months; colonoscopy within 10 years; sigmoidoscopy within 5 years; barium enema within 5 years, CT colonography within 10 years

Ages: 52 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2144 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Number of participants who completed fecal testing, screening colonoscopy, and colonoscopies following positive fecal testing, • | 21 months following baseline
  Screening status will be assessed through participant response and Medicaid claim data.
Diagnoses of colorectal Cancer | 21 months following baseline
  Diagnoses of colorectal cancer will be assessed through Medicaid claim data.
Polypectomies | 21 months following baseline
  Number of polypectomies will be assessed through Medicaid claim data.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Brenner, PhD, MPH, Principal Investigator — UNC Lineberger Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No